CLINICAL TRIAL: NCT01445015
Title: Pilot Study: Stress Management Intervention as a Tool for Managing Persistent Asthma in Inner City Adolescent Patients.
Brief Title: Stress Management Intervention in Inner City Adolescents With Asthma
Acronym: SIPIICAA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Lisa Moreno, MD, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5T32HS000066 (AHRQ)
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Asthma; Psychosocial Stress
Keywords: adolescents
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress management program (Experimental)
  Interventions: Behavioral: Stress management program
- peer viewed movies (Active Comparator)
  Interventions: Other: Peer viewed movies

INTERVENTIONS:
Behavioral: Stress management program — 10 session intervention utilizing a cognitive behavorial program with a goal of stress reduction
  Arms: Stress management program
Other: Peer viewed movies — PG rated movies to be viewed over 10 sessions in peer setting
  Arms: peer viewed movies

SUMMARY:
The study will utilize a stress management program delivered over 10 sessions that is hypothesized to result in decreased stress levels and improved coping strategies in an inner city adolescent asthma population. Participants will include adolescents ages 10-15 years with physician diagnosed asthma. The outcome measures will be obtained via psychosocial questionnaires and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-15 years of age
* Physician diagnosed asthma based on NHBLI guidelines
* English speaking
* Child assent/parental consent

Exclusion Criteria:

* Refusal of child assent/parental consent
* Non-English speaking
* History of psychiatric illness, autoimmune disease, HIV/AIDs, smoking history.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-02 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Scope of change in perceived stress from enrollment to completion of study using the Perceived stress scale | 5 weeks

SECONDARY OUTCOMES:
Secondary outcomes within scope of change from enrollment to completion of study in coping as assessed by Kidcope | 5 weeks
Secondary outcomes within scope of change from enrollment to completion of study in anxiety as measured by State Trait Inventory | 5 weeks
Secondary outcomes within scope of change from enrollment to completion of study in quality of life as assessed by PAQLQ | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell Weill Pulmonary/Allergy pediatric clinics, New York, New York, United States